CLINICAL TRIAL: NCT00638352
Title: Determination of the False Negative Rate of Percutaneous Needle Biopsies That Include Core Tissue Samples
Brief Title: False/Negative Rate of Lung Percutaneous Needle Biopsy
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Ernest Scalzetti, MD, State University of New York - Upstate Medical University
Other Study IDs: SUNYUMU 5334
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Lung Neoplasm
Keywords: Core Biopsy; Needle Biopsy; Percutaneous Biopsy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Needle biopsy is a way of determining whether a lung mass is cancerous or benign. Its accuracy was established by research in which patients underwent fine needle aspiration, a kind of needle biopsy that yields samples for cytology (similar to the way a pap smear or a fluid sample would be evaluated for malignant cells). This kind of needle biopsy may supplemented or replaced by core needle biopsy, which yields samples for histology (similar to surgical tissue samples but on a smaller scale) rather than for cytology. Core needle biopsy is believed to be helpful particularly in obtaining a diagnosis in patients who have a lung mass that their doctors think is cancerous but is, in fact, benign. In spite of the advances in needle biopsy, however, there are patients who do receive a pathology report indicating no evidence of cancer but whose lung mass actually is cancerous. The fraction of such patients, among all patients who have no evidence of cancer according to the biopsy, is called the "false negative rate." It is approximately 25% for needle biopsies that consist of fine needle aspiration alone. The false negative rate for needle biopsies that include core biopsy samples is not known.

We want to examine the accuracy of needle biopsy in patients who had core samples taken from a lung mass in addition to, or in place of, fine needle aspiration. In this study we will focus on such patients who had no evidence of cancer according to the biopsy, to determine how many actually had a cancer that was missed by the biopsy. To accomplish this goal, we will need to review the medical records of these patients for one of two things: either a definitive diagnosis of the lung mass by some other means (for example, surgical biopsy), or by seeing how the patient does over a period of time (usually in conjunction with medical imaging tests such as chest x-rays or chest CT scans). To establish that a lung mass is benign by observing a patient over time, it is necessary to show that the lung mass disappears, becomes smaller, or remains unchanged in size for 2 years.

DETAILED DESCRIPTION:
We will review medical records to identify patients who underwent percutaneous needle biopsy of a lung mass between 5/1/01 and 10/30/04. If the pathology report indicates that the biopsy showed no evidence of malignancy, we will examine the medical record for a "gold standard" diagnosis of the lesion in question, including the pathology result from a surgical resection or a repeat biopsy, imaging follow-up demonstrating regression of the lesion or size stability for at least 2 years, or clinical follow-up for at least 2 years with no clinical evidence of malignant disease. If this information is not available in the University Hospital medical record, we will contact the patient to obtain consent for follow-up using external sources (physician records, imaging studies, pathology reports).

We will derive descriptive statistics (prevalence of malignancy, sensitivity, specificity, and false negative rates). The overall sample size will be ~500 patients who had PTNB of a lung mass within the study period. Approximately 80 are expected to have a biopsy result showing no evidence of malignancy, based on a retrospective review performed under an IRB exemption (87-04, letter dated 9/28/04). The expected proportion of cases with no evidence of malignancy is approximately 0.15. For a 95% confidence interval of 0.15+/-0.075 we will need follow-up information from 61 patients, considering that this is a descriptive study with a dichotomous variable. This gives us a margin for patients who will be lost to follow-up

ELIGIBILITY:
Inclusion Criteria:

* subjects who underwent percutaneous needle biopsy of a lung mass during the study period of 5/1/01 to 10/30/04

Exclusion Criteria:

* subjects will be excluded if at least one core sample was not obtained in the course of the biopsy.
* subjects who had a pathology sample read as "insufficient for diagnosis"
* subjects who underwent needle biopsy only for infection, to identify a causative organism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will review medical records to identify patients who underwent percutaneous needle biopsy of a lung mass between 5/1/01 and 10/30/04. If the pathology report indicates that the the biopsy showed no evidence of malignancy, we will examine the medical record for a "gold standard" diagnosis of the lesion in question, including the pathology result from a surgical resection or a repeat biopsy, or imaging follow-up demonstrating regression of the lesion (or size stability for at least 2 years), or clinical follow-up for at least 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine the false negative rate of PTNB procedures that include core tissue samples, and to compare it to the historical false negative rate of PTNB with FNA only. | 2 years

SECONDARY OUTCOMES:
To determine the sensitivity of PTNB procedures that include at least one core tissue sample, for the diagnosis of malignancy. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Scalzetti, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No